CLINICAL TRIAL: NCT04288895
Title: Open-label, Flexible-dose Study of Vortioxetine in Patients With Major Depressive Disorder in India
Brief Title: Open-label, Flexible-dose Study of Vortioxetine in Patients With Depression in India
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17775A
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vortioxetine (Experimental): flexible-dose
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — 5 - 20 mg/day flexible-dose vortioxetine, tablets, orally

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of flexible doses of vortioxetine (5 - 20 mg/day) over a period of 12 weeks in patients with depression in India

ELIGIBILITY:
Inclusion Criteria:

* The patient has a Major Depressive Episode (MDE), is diagnosed with Major Depressive Disorder (MDD) according to DSM-5® and would benefit from pharmacological treatment with vortioxetine. The current MDE should be confirmed using the Mini International Neuropsychiatric Interview (MINI).
* The patient has a CGI-S ≥4 at screening.

Exclusion Criteria:

* The patient has a significant risk of suicide according to investigator's clinical judgment or has made an actual suicide attempt in the period of 6 months prior to screening.
* The patient previously received vortioxetine.

Other in- and exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-03-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment-Emergent Adverse Events | From baseline to week 12

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) total score | From baseline to week 12
  The PHQ-9 is a patient-rated scale designed to screen for and assess depression. The PHQ-9 consists of questions on each of the 9 DSM-5® criteria for depression asking if they have bothered the patient over the last 2 weeks. Each question is rated on a scale from 0 (not at all) to 3 (nearly every day). The 9 questions are summed to a total score ranging from 0 to 27 with higher scores reflecting greater severity.
Change in Clinical Global Impression-severity of illness (CGI-S) score | From baseline to week 12
  The CGI was developed to provide global measures of the severity of a patient's clinical condition and improvement or worsening during clinical studies. The CGI consists of two clinician-rated subscales: severity of illness (CGI-S) and global improvement (CGI-I). The CGI-S provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill patients).
Clinical Global Impression-improvement (CGI-I) | At week 12
  The CGI was developed to provide global measures of the severity of a patient's clinical condition and improvement or worsening during clinical studies. The CGI consists of two clinician-rated subscales: severity of illness (CGI-S) and global improvement (CGI-I). The CGI-I provides the clinician's impression of the patient's improvement (or worsening). The clinician assesses the patient's condition relative to a baseline on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse).

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (24):
- India (24):
  - Ratandeep Multispecialty Hospital (IN1002), Ahmedabad, Gujarat
  - MITR Foundation 1 (IN1013), Ahmedabad, Gujarat
  - BJ Medical College and Civil Hospital (IN028), Ahmedabad, Gujarat
  - Shree Hatkesh Health Foundation (IN1016), Jūnāgadh, Gujarat
  - Nagecha Hospital, Creative Chamber (IN1015), Rajkot, Gujarat
  - Divyam Clinic (IN1025), Surat, Gujarat
  - GMERS Medical College and Hospital,Department of Psychiatry (IN1004), Vadodara, Gujarat
  - People Tree Hospitals (IN1027), Bengaluru, Karnataka
  - Vinaya Hospital & Research Centre (IN1007), Mangalore, Karnataka
  - Mangala Hospital & Mangala Kidney Foundation (IN1006), Mangalore, Karnataka
  - K. S. Hegde Medical Academy (IN1003), Mangalore, Karnataka
  - Department of Psychiatry K R Hospital Mysore Medical College and Research Institute (IN1020), Mysuru, Karnataka
  - IQRAA International Hospital & Research Centre (IN030), Kozhikode, Kerala
  - Society for Psychiatric Update and Research, Shanti Nursing Home (IN1008), Aurangabad, Maharashtra
  - Arneja Heart and Multispeciality Hospital (IN1022), Nagpur, Maharashtra
  - Central Institute of Behavioural Sciences (IN1019), Nagpur, Maharashtra
  - Chopda Medicare & Research Centre (IN023), Nashik, Maharashtra
  - Lata Mangeshkar Medical Foundation's (IN1001), Pune, Maharashtra
  - Oyster and Pearl Hospital (IN1014), Pune, Maharashtra
  - Dayanand Medical College and Hospital (IN024), Ludhiana, Punjab
  - ASHA hospital (IN1018), Hyderabad, Telangana
  - Deva Institute of Healthcare and Research PVT ltd. (IN1005), Varanasi, Uttar Pradesh
  - Institute of Post Graduate Medical Education and Research (IN1026), Kolkata, West Bengal
  - Maharaja Agarsen Hospital (IN1021), Delhi

REFERENCES:
- [Derived] Adair M, Bose R, Schmidt SN. Safety and effectiveness of vortioxetine in patients with major depressive disorder in a real-life clinical setting in India: results from an interventional, flexible-dose study. Curr Med Res Opin. 2024 Sep;40(9):1637-1645. doi: 10.1080/03007995.2024.2382773. Epub 2024 Aug 7. PMID 39110846